CLINICAL TRIAL: NCT02384330
Title: Cost Determination Study For Different Botulinum Toxin A Preparations In The Treatment Of Upper Limb Spasticity Post-Stroke In Portugal
Brief Title: Botulinum Toxin A Associated Costs in the Treatment of Upper Limb Spasticity Post Stroke
Acronym: P_Dysport_CS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52120-188
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Upper Limb Spasticity Post-Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Dysport® (abobotulinumtoxinA): Botulinum Toxin Type A (BoNT-A) preparation, injected doses, number of points, volume per point, in accordance with local Summary of Product Characteristics and locally agreed therapeutic guidelines.
- Botox® (onabotulinumtoxinA): Botulinum Toxin Type A (BoNT-A) preparation, injected doses, number of points, volume per point, in accordance with local Summary of Product Characteristics and locally agreed therapeutic guidelines.
- Xeomin® (incobotulinumtoxinA): Botulinum Toxin Type A (BoNT-A) preparation, injected doses, number of points, volume per point, in accordance with local Summary of Product Characteristics and locally agreed therapeutic guidelines.

SUMMARY:
This study aims to estimate the costs of botulinum toxin A utilization in standard practice for the treatment of upper limb spasticity post-stroke in Portugal.

It will consider the three most used locally available brands of botulinum toxin A which show similar efficacy and safety profiles thus making it relevant to understand if choosing between one or another brand can depend directly on economic factors.

The study will estimate direct and indirect drug-associated costs as determinant variables for the price of each drug and the standard drug dose used in clinical practice.

DETAILED DESCRIPTION:
A comparison will be performed between direct costs associated with each therapeutic strategy and cost analysis assuming that quality of life values may be different between patients treated with each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with post-stroke upper limb spasticity
* Patients currently being treated with Dysport®, Botox® or Xeomin®
* Patients stabilized from a therapeutic point of view - with no switches of treatment in at least the 2 last administrations
* Patients who gave their written informed consent to participate.

Exclusion Criteria:

* Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital ambulatory patients
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Estimate the cost of botulinum toxin utilization | 12 months
  Direct resource utilization and costs of upper limb spasticity patients treated with BoNT-As, by product

SECONDARY OUTCOMES:
Number of work days missed due to spasticity | 12 months
  Assessment of Absenteeism /loss of productivity
Carer time needed for patient assistance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- Portugal (3):
  - Centro de Medicina de Reabilitação de Alcoitão, Alcabideche
  - C. H. A. - Hospital de Faro, Faro
  - C. H. T. M. A. D. - Unidade Hospitalar de Vila Real, Vila Real